CLINICAL TRIAL: NCT04453956
Title: A Prospective, Randomized, Single-blind, 2 × 2 Factorial Design Single Center Study Evaluating the Polyp Detection and Quality Monitoring Function of EndoAngel in Improving the Quality of Colonoscopy
Brief Title: A Single Center Study on Comparing the Different Function of EndoAngel in Improving the Quality of Colonscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: EA-19-001
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Adenoma
Keywords: Polyp Detection; Quality Monitoring; Artificial Intelligence
MeSH Terms: conditions — Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Sham Comparator): Patients will receive colonoscopy without assistance of EndoAngel's any function.
  Interventions: Diagnostic Test: Colonoscopy without the assistance of EndoAngel's any function.
- Polyp detection function group (Experimental): Patients will receive colonoscopy with the assistance of EndoAngel's polyp detection function.
  Interventions: Diagnostic Test: Colonoscopy with the assistance of EndoAngel's polyp detection function.
- Quality monitoring function group (Experimental): Patients will receive colonoscopy with the assistance of EndoAngel's quality monitoring function.
  Interventions: Diagnostic Test: Colonoscopy with the assistance of EndoAngel's quality monitoring function.
- Polyp detection plus quality monitoring functions group (Experimental): Patients will receive colonoscopy with the assistance of EndoAngel's polyp detection plus quality monitoring function.
  Interventions: Diagnostic Test: Colonoscopy with the assistance of EndoAngel's polyp detection function.; Diagnostic Test: Colonoscopy with the assistance of EndoAngel's quality monitoring function.

INTERVENTIONS:
Diagnostic Test: Colonoscopy with the assistance of EndoAngel's polyp detection function. — Patient in this group will receive colonoscopy with assistance of EndoAngel's polyp detection function,which can remind endoscopists of the location of the polyp.
  Arms: Polyp detection function group; Polyp detection plus quality monitoring functions group
Diagnostic Test: Colonoscopy with the assistance of EndoAngel's quality monitoring function. — Patient in this group will receive colonoscopy with assistance of EndoAngel's quality monitoring function,which can monitor the withdrawal speed of the endoscope.
  Arms: Polyp detection plus quality monitoring functions group; Quality monitoring function group
Diagnostic Test: Colonoscopy without the assistance of EndoAngel's any function. — Patient in this group will receive colonoscopy with assistance of EndoAngel's both functions.
  Arms: Control group

SUMMARY:
An artificial intelligence-based system, named EndoAngel,has been constructed previously,which has polyp detection and quality monitoring functions. This study aims to evaluate the two different functions of EndoAngle in improving adenoma detection rate.

DETAILED DESCRIPTION:
The detection and removal of precancerous polyps via colonoscopy can reduce the the risk of colon cancer. However, the detection rate of adenomatous polyps can vary significantly among endoscopists. EndoAngel is an artificial intelligence-based system,consisting of polyp detection and quality monitoring functions. The polyp detection function can remind endoscopists of the location of the polyp. The quality monitoring function can monitor the velocity of insertion of the endoscope, record the time of insertion and withdrawal of the endoscope, and remind endoscopists of the blind areas caused by intestinal segment slipping.This study aims to evaluate the two different functions of EndoAngle by 2 × 2 factorial design in improving adenoma detection rate and the quality of colonscopy .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or above;
2. Colonoscopy is needed to further characterize gastrointestinal diseases;
3. Ability to read, understand and sign informed consent forms;
4. The researchers believe that the subjects can understand the process of the clinical study and are willing and able to complete all the study procedures and follow-up visits to cooperate with the study procedures.

Exclusion Criteria:

1. Participated in other clinical trials, signed informed consent forms and followed up in other clinical trials；
2. Participate in a drug clinical trial and during the elution period of the trial or control drug；
3. Drug or alcohol abuse or mental disorder in the last 5 years;
4. Pregnant or lactating women;
5. Patients with multiple polyp syndrome;
6. Patients with a history of inflammatory bowel disease, colorectal cancer, or colorectal surgery;
7. Patients with known perforation or colonic obstruction;
8. Patients with a contraindication for biopsy;
9. The researchers did not consider the subjects suitable for colonoscopy;
10. The researchers determined that the subjects had high-risk diseases or other special conditions that were not appropriate for clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1090 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-20 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 3 Months
  The numerator is the number of cases of adenomas detected by colonoscopy, and the denominator is the total number of cases of patients undergoing colonoscopy.

SECONDARY OUTCOMES:
Polyp detection rate | 3 months
  The numerator is the number of cases of polyps detected by colonoscopy, and the denominator is the total number of cases of patients undergoing colonoscopy.
The mean number of polyps per procedure | 3 months
  The numerator is the total number of polyps detected by colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
The mean number of adenomas per procedure | 3 months
  The numerator is the total number of adenomas detected by colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
Detection rate of large, small and diminutive polyps | 3 months
  The numerator was the number of patients with large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
The mean number of large, small and diminutive polyps per procedure | 3 months
  The numerator was the number of large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
Detection rate of large, small and diminutive adenomas | 3 months
  The numerator was the number of patients with large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) adenomas detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
The mean number of large, small and diminutive adenomas per procedure | 3 months
  The numerator was the number of large (≥10 mm), small (>5 to <10 mm), and diminutive(≤5 mm) adenomas detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
Detection rate of adenoma in different sites | 3 months
  The numerator is the number of cases of adenoma detected in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon and ileocecal region during colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
The mean number of adenomas in different sites per procedure | 3 months
  The numerator is the total number of adenomas detected in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon and ileocecal region during colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
Time of colonoscopic insertion | 3 months
  The duration of colonoscopic insertion from rectum to ileocecal valve or appendiceal opening
Time of colonoscopic withdrawal | 3 months
  The duration of colonoscopic withdrawal from ileocecal valve or appendiceal opening to colonoscopy finished.
Cecal intubation rate | 3 months
  The numerator is the number of cases of colonoscopy reaching ileocecal valve or appendiceal opening, and the denominator is the total number of colonoscopy cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yao L, Zhang L, Liu J, Zhou W, He C, Zhang J, Wu L, Wang H, Xu Y, Gong D, Xu M, Li X, Bai Y, Gong R, Sharma P, Yu H. Effect of an artificial intelligence-based quality improvement system on efficacy of a computer-aided detection system in colonoscopy: a four-group parallel study. Endoscopy. 2022 Aug;54(8):757-768. doi: 10.1055/a-1706-6174. Epub 2022 Feb 4. PMID 34823258